CLINICAL TRIAL: NCT03544151
Title: Swan-Ganz CCOmbo V for Obtaining an Optimal Depth of Right Internal Jugular Venous Catheter : A Prospective Observational Study
Brief Title: Swan-Ganz CCOmbo V for Obtaining an Optimal Depth of Right Internal Jugular Venous Catheter
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-012
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Insertion Depth of Central Venous Catheter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Swan-Ganz Continuous Cardiac Output Thermodilutioon Cather (Swan-Ganz CCOmbo V) — Swan-Ganz CCOmbo V insertion

SUMMARY:
The investigators will perform a study to create formula for the optimal insertion depth of right internal jugular vein catheter.

DETAILED DESCRIPTION:
Patients scheduled for cardiac surgery were studied.Determine the optimal insertion depth of right internal jugular vein catheter using Swan-Ganz Continuous Cardiac Output Thermodilutioon Cather (Swan-Ganz CCOmbo V).The investigators measure the distance between the insertion point and the junction between right atrium and superior vena cava using Swan-Ganz CCOmbo V.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient over 18 years of age undergoing mitral valve or/and tricuspid valve
* Surgery under general anesthesia, requiring Swan-Ganz Continuous Cardiac Output Thermodilutioon Cather (Swan-Ganz CCOmbo V) insertion through the right internal jugular vein.

Exclusion Criteria:

* A change in the mediastinal structure from previous neck surgery,thoracic surgery or cardiac surgery
* Extracardiac vascular anomaly
* Anatomical abnormality in neck and thorax
* Refusal to enrol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for cardiac surgery were studied
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-12-27 (Actual)

PRIMARY OUTCOMES:
The distance | After insertion of the Swan-Ganz Continuous Cardiac Output Thermodilutioon Cather (Swan-Ganz CCOmbo V) and during operation
  The distance between the insertion point and the junction between right atrium and superior vena cava

CONTACTS AND LOCATIONS:
Overall Officials: qi lu, Dr., Study Director — Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China
Locations (1):
- Diansan Su, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided